CLINICAL TRIAL: NCT07390188
Title: Prevalence of Oral Mucosal Lesions Among a Sample of Adult Egyptian Subjects: Hospital Based Cross-sectional Study.
Brief Title: Prevalence of Oral Mucosal Lesions Among a Sample of Adult Egyptian Subjects
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eslam EL Sayed Abdelfattah El Zayat, Master's Candidate, Cairo University
Other Study IDs: OMED 1.1.1
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucosal Disease; Oral Mucosal Disorder
Keywords: Oral Mucosal Lesions; OML; OMLs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral mucosal lesion represents a wide array of conditions. They may be the result of a local or systemic infection or trauma or the manifestations of a medical condition or neoplastic growth weather primary or metastatic or may be mistaken for a variation of a normal structure. This study aims to estimate the prevalence of OMLs and describe the risk factors for the development of OMLs in a sample of the Egyptian population Research Question :What is the prevalence of oral mucosal lesions and their associated risk factors in a sample of adult Egyptians?

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years old and above, Egyptian individuals

Exclusion Criteria:

* Individuals refusing to participate in the study. Individuals unable to give accurate or full information due to suffering from acute symptoms, requiring immediate intervention. Individuals unable to give accurate or full information due to any disease preventing them from opening their mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals, above 18 years old, presenting for initial diagnosis to DC of outpatient clinic of Faculty of Dentistry, Cairo university.
Sampling Method: Non-Probability Sample
Enrollment: 14645 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Lesion Presence | At Time of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt